CLINICAL TRIAL: NCT01097915
Title: Sensitivity to 6-n-propylthiouracil (PROP) Association With Gustin (CA6) Gene Polymorphism, Salivary Zinc and BMI in Humans
Brief Title: Gustin Gene Polymorphism and 6-n-propylthiouracil (PROP) Taste
Acronym: gustinprop
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Iole Tomassini Barbarossa, Associate Professor, University of Cagliari
Other Study IDs: UNICADBSITB-1
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Dysgeusia
Keywords: PROP taste sensitivity; Gustin (CAVI) polymorphism; Salivary zinc; BMI; Electrophysiological recording from the tongue
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and zinc analyses in saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROP taste sensitivity: PROP Sensitive and non sensitive individuals are defined as "Tasters" and "Non-tasters", respectively. Taster are further divided in "Super-taster" who perceived PROP as extremely bitter and "Medium tasters" who perceived PROP as moderately bitter.

SUMMARY:
The investigators evaluate the possible association of PROP taste with gustin gene polymorphism rs2274333 (A/G), salivary zinc ion concentration and BMI. In addition, it has also been evaluated PROP taste sensitivity by recording monophasic potentials from the tongue.

DETAILED DESCRIPTION:
The investigators evaluate the possible association of PROP taste with gustin gene polymorphism rs2274333 (A/G), salivary zinc ion concentration and BMI.

Furthermore, we apply direct measures of the gustatory system activation following stimulation with PROP, obtained by electrophysiological recordings from the tongue of subjects classified for taster status, genotyped for the specific receptor gene (TAS2R38), and in which papilla density was determined.

ELIGIBILITY:
Inclusion Criteria:

* no variation of body weight > 5 kg over the last 3 mo BMI within 20-25 Age between 20-30

Exclusion Criteria:

* gustatory impairment following a prescribed diet or using medications that might interfere with taste perception food allergies smokers

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Seventy-five non-smoking volunteers (28 men and 47 women) were recruited for the study. Participants between 20-30 years were eligible for the study. Thresholds for the 4 basic tastes were evaluated in all subjects in order to rule out any gustatory impairment. The volunteers showed no variation of body weight > 5 kg over the last 3 mo. They were not following a prescribed diet or using medications that might interfere with taste perception; none had food allergies. They were assessed for cognitive eating behaviours using the Three-Factor Eating Questionnaire
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iole Tomassini Barbarossa, PhD, Principal Investigator — Dip. Scienze Biomediche Sezione di Fisiologia Università di Cagliari
Locations (1):
- Sezione di Farmacologia Clinica del Dipartimento di Neuroscienze, San Giovanni di Dio Azienda Ospedaliero Universitaria di Cagliari, Cagliari, Ca, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data of this study are available from the principal investigator of this study upon request

REFERENCES:
- [Derived] Padiglia A, Zonza A, Atzori E, Chillotti C, Calo C, Tepper BJ, Barbarossa IT. Sensitivity to 6-n-propylthiouracil is associated with gustin (carbonic anhydrase VI) gene polymorphism, salivary zinc, and body mass index in humans. Am J Clin Nutr. 2010 Sep;92(3):539-45. doi: 10.3945/ajcn.2010.29418. Epub 2010 Jul 14. PMID 20631203

RESULTS

PARTICIPANT FLOW:
Groups:
- Super Tasters: Subjects highly sensitive to PROP
- Medium Tasters: Subjects sensitive to PROP
- Non Tasters: Subjects no sensitive to PROP
Period: Overall Study
Arm/Group | Super Tasters | Medium Tasters | Non Tasters
Started | 50 | 70 | 50
Completed | 27 | 28 | 20
Not Completed | 23 | 42 | 30

BASELINE CHARACTERISTICS:
Population: Caucasian and were originally from Sardinia, Italy. Participants between 20-30 years were eligible for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Super Tasters | Medium Tasters | Non Tasters | Total
Number analyzed (Participants) | 50 | 70 | 50 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 70 | 50 | 170
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (7) | 25 (8) | 25 (6) | 25 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 34 | 109
  Male | 15 | 30 | 16 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 50 | 70 | 50 | 170
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 50 | 70 | 50 | 170
healthy volunteers [Number; unit: participants] | 50 | 70 | 50 | 170

OUTCOME MEASURES:

1. Primary Outcome: Association Between Gustin Gene Polymorphism and PROP Sensitivity
Description: We examine associations between PROP status and the polymorphism rs2274333 (A/G) of the gene that codify for the salivary protein, gustin/CA6, Which has been suggested as a trophic factor that promotes growth and development of taste buds by acting on taste bud stem cells.
  The intensity of taste perception evoked by PROP and NaCl solutions was estimated to evaluate PROP taster status and molecular analysis of the gustin gene polymorphism was performed in individuals classified by PROP status using PCR techniques.
Time Frame: 7 months
Measure: Number; unit: percentage of participants
Arm/Group | Super Tasters | Medium Tasters | Non Tasters
Number analyzed (Participants) | 27 | 28 | 20
percentage of participants
  Genotype AA | 85.19 | 50.99 | 25.00
  Genotype AG | 14.81 | 35.71 | 20
  Genotype GG | 0 | 14.29 | 55
  Allele A | 92.59 | 67.86 | 35
  Allele G | 7.40 | 32.14 | 65
Statistical Analysis 1: Comparison: Super Tasters vs Medium Tasters vs Non Tasters; Test type: Superiority or Other; p < 0.01, Fisher Exact

2. Secondary Outcome: Association Between PROP Sensitivity and Saliva Zinc Ion Concentration
Description: Since the enzymatic function of gustin (CA6) depends upon the presence of Zn at its active site we measured the salivary zinc ion concentration in subjects classified as super-taster, medium taster and non-taster.The salivary Zn2+ concentration was measured with a QuantiChromTM zinc Assay kit (Gentaur, Brussels, Belgium) where the color intensity is directly proportional to the Zn2+ concentration in the sample.
Time Frame: 7 months
Measure: Mean (Standard Error); unit: microg/dl
Groups:
- Super-tasters: Subjects highly sensitive to PROP
- Non-tasters: Subjects no sensitive to PROP
Arm/Group | Super-tasters | Medium Tasters | Non-tasters
Number analyzed (Participants) | 27 | 28 | 20
microg/dl | 57.3 (13) | 89.5 (17.2) | 149.64 (26.4)
Statistical Analysis 1: Comparison: Super-tasters vs Medium Tasters vs Non-tasters; Test type: Superiority or Other; p < 0.004, ANOVA

3. Secondary Outcome: Association Between PROP Sensitivity and BMI
Description: Since individual ability to taste PROP may be correlated with BMI, we determined BMI (kg/m^2) in subjects classified as super-taster, medium taster and non-taster.Weight (kg) and height (m) were recorded for each subject.
Time Frame: 7 months
Measure: Mean (Standard Error); unit: Kg/m^2
Arm/Group | Super-tasters | Medium Tasters | Non-tasters
Number analyzed (Participants) | 27 | 28 | 20
Kg/m^2 | 20.3 (0.48) | 20.76 (0.58) | 22.58 (0.84)
Statistical Analysis 1: Comparison: Super-tasters vs Medium Tasters vs Non-tasters; Test type: Superiority or Other; p < 0.048, ANCOVA; the three factors of the Stunkard and Messick Questionnaire were considered as covariates

4. Secondary Outcome: Electrophysiological Recordings From the Tongue for the Objective Evaluation of Individual Variations of 6-n-propylthiouracil (PROP) Sensitivity
Description: electrophysiological recordings from the tongue of 43 subjects classified for their taste sensitivity to 6-n- propyltiouracil (PROP) and genotyped for the specific receptor gene, TAS2R38. Density of fungiform papillae was also determined in each subject. The biopotentials were recorded by means of differential electrophysiological derivations between two silver electrodes, one in contact with the ventral surface of the tongue and one in perfect adhesion with the dorsal surface.
Time Frame: 1 year
Population: Relationship between depolarization amplitude of signals and PROP taster status.
Measure: Mean (Standard Error); unit: mV
Groups:
- Super-Taster: Subjects highly sensitive to PROP
- Medium Taster: Subjects sentitive to PROP
- Non Taster: Subjects no sensitive to PROP
Arm/Group | Super-Taster | Medium Taster | Non Taster
Number analyzed (Participants) | 15 | 15 | 13
mV | 97,08867 (6,538191) | 75,42000 (6,538191) | 48,48231 (7,023144)
Statistical Analysis 1: Comparison: Super-Taster vs Medium Taster vs Non Taster; Test type: Superiority or Other; p < 0.00001, ANOVA

5. Secondary Outcome: Association Between PROP Sensitivity and Fungiform Papilla Density
Description: 43 subjects were classified for their taste sensitivity to 6-n- propyltiouracil (PROP) and density of fungiform papillae was determined in each subject.
Time Frame: 6 months
Population: Relationship between density of fungiform papillae and PROP taster status.
Measure: Mean (Standard Error); unit: No./cm2
Arm/Group | Super-tasters | Medium Tasters | Non-tasters
Number analyzed (Participants) | 15 | 15 | 13
No./cm2 | 51.66 (5.25) | 33.49 (5.26) | 18.53 (7.023)
Statistical Analysis 1: Comparison: Super-tasters vs Medium Tasters vs Non-tasters; Test type: Superiority or Other; p < 0.00001, ANOVA

6. Secondary Outcome: Taste Perception of Sweet, Sour, Salty, Bitter and Umami and Changes Due to L-Arginine Supplementation, as a Functin of Genetic Ability to Taste PROP.
Description: Taste perception was assessed by testing the ability to recognize, and the responsiveness to, representative solutions of the five taste qualities, also when supplemented with L-Arg, in subjects classified as PROP-tasters.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- Primary Taste Quality: we taste Sucrose, NaCl, Citric Acid, Caffeine and MSG
- Primary Taste Quality Supplemented With L-Arg: we taste Sucrose, NaCl, Citric Acid, Caffeine and MSG, each supplemented with L-Arginine (1:1)
Arm/Group | Primary Taste Quality | Primary Taste Quality Supplemented With L-Arg
Number analyzed (Participants) | 64 | 64
Participants
  sucrose: Undet Threshold | 18 | 2
  sucrose: Correct identification | 40 | 20
  sucrose: Incorrect teste response | 6 | 42
  NaCl: Undet Threshold | 1 | 1
  NaCl: Correct identification | 52 | 41
  NaCl: Incorrect teste response | 11 | 22
  Citric Acid: Undet Threshold | 5 | 4
  Citric Acid: Correct identification | 49 | 47
  Citric Acid: Incorrect teste response | 10 | 13
  caffeine: Undet Threshold | 6 | 6
  caffeine: Correct identification | 56 | 56
  caffeine: Incorrect teste response | 2 | 2
  MSG: Undet Threshold | 7 | 0
  MSG: Correct identification | 26 | 33
  MSG: Incorrect teste response | 31 | 31
Statistical Analysis 1: Comparison: Primary Taste Quality vs Primary Taste Quality Supplemented With L-Arg; Test type: Superiority or Other; p < 0.00001, Chi-squared

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Super Tasters | Medium Tasters | Non Tasters
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/20
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No